CLINICAL TRIAL: NCT05979740
Title: RC48 Combined With PD-1 and Radiotherapy as Bladdersparing Therapy in Patients With Muscular Infiltrating Bladder Uroepithelial Carcinoma With Limited HER-2 Expression Following Maximum Electrical Resection or Partial Cystectomy
Brief Title: RC48 Combined With Toripalimab and Radiotherapy for Bladder Sparing Treatment in MIBC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2023-002-A
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Muscle Invasive Bladder Cancer; HER2 Expression; Radiotherapy; PD-1; Antibody-drug Conjugates
Keywords: Muscle Invasive Bladder Cancer; HER2 expression; Radiotherapy; PD-1; ADC; Bladder Sparing
MeSH Terms: interventions — disitamab vedotin; toripalimab; RC48 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48+Toripalimab+Radiotherapy (Experimental): RC48: 2.0 mg/kg, Q2W, iv; Toripalimab: 3mg/kg, Q2W, iv; Radiotherapy: total dose was greater than 50Gy (about 30 times).
  Interventions: Drug: Disitamab Vedotin and Toripalimab

INTERVENTIONS:
Drug: Disitamab Vedotin and Toripalimab — Each patient received RC48 injection [2.0 mg/kg, Q2W, iv] and Toripalimab injection [3mg/kg, Q2W, iv] for 1~2 cycles, and Radiotherapy radiotherapy at the second or third cycle. The total dose of bladder irradiation field was greater than 50Gy (about 30 times), and the safety monitoring of the subjects was conducted within 28 days after receiving the study drug treatment for the first time.
  Other Names: RC48, JS001

SUMMARY:
This is a prospective, open, single-center clinical study of RC48 combined with PD-1 and radiotherapy as bladder-preserving therapy in patients with muscular invasive bladder uroepithelial carcinoma with high HER-2 expression (IHC 2+ or 3+). The study was conducted in accordance with the Good Practice for Clinical Trials of Pharmaceutical Products (GCP). Six patients were enrolled in this study. Each patient received RC48 injection [2.0 mg/kg, Q2W, iv] and Toripalimab injection [3mg/kg, Q2W, iv] for 1~2 cycles, and radiotherapy at the second or third cycle. The total dose of bladder irradiation field was greater than 50Gy (about 30 times), and the safety monitoring of the subjects was conducted within 28 days after receiving the study drug treatment for the first time. Adverse events were graded using the National Cancer Institute (NCI) Standard for the Assessment of Common Terminology for Adverse Events (CTCAE) Version 5.0 guidelines, and the occurrence of DLT in patients was observed. If the subject does not complete the safety assessment for the tolerance observation period for non-dose tolerance reasons, a new subject will be replaced.

DETAILED DESCRIPTION:
This is a prospective, open, single-center clinical study of RC48 in combination with PD-1 and radiotherapy as bladder-preserving therapy in patients with muscular invasive bladder uroepithelial carcinoma with high HER-2 expression (IHC 2+ or 3+). The study was conducted in accordance with the Good Practice for Clinical Trials of Pharmaceutical Products (GCP).

Subjects undergo maximum transurethral electrocystotomy (TURBT) or partial cystectomy, imaging diagnosis, and pre-treatment biological samples of blood, urine, and biopsy tissue. The researchers determined that localized invasive bladder cancer with high HER-2 expression could be treated with bladder conserving therapy with maximum TURBT. Patients will receive RC48 combined with PD-1 and radiotherapy after TURBT surgery. Subjects should receive RC48 combined with PD-1 every two weeks for 12 treatment cycles and radiotherapy (bladder irradiation field greater than 50Gy). After completion of the above treatment, tumor site pathology, imaging, and exfoliation cytology are obtained with diagnostic TURBT for tumor evaluation to determine complete remission, and the first tumor efficacy evaluation is performed after completion of radiotherapy (12 weeks after treatment) and every 12 weeks after completion of radiotherapy. Patients with radiotherapy intolerance (as assessed by the investigator) were discontinued directly.

Adverse events will be monitored during the study period and graded using the National Cancer Institute's (NCI) Standards for the Assessment of Adverse Events in General Terminology (CTCAE) Version 5.0 guidelines. The safety assessment was carried out after 28 days.

Subjects who discontinue medication for reasons other than disease progression will be followed for post-treatment disease status until subjects begin other antitumor therapy, develop disease progression, withdraw informed consent, die, or end of the study, whichever occurs first. All subjects will be followed up via outpatient cystoscopy (every 3 months within 1 year of withdrawal and every 6 months after 1 year) until subject's death, withdrawal of informed consent, or the end of the study, whichever occurs first.

Participation in this study will require participants to submit a TURBT tumor tissue specimen or a newly obtained tumor lesion biopsy from prior untreated radiation therapy for biomarker and efficacy correlation evaluation.

Blood and urine samples from patients will be collected during the treatment to explore potential biomarkers correlated to the treatment efficacy and patient response.

ELIGIBILITY:
Inclusion criteria:

ECOG PS: 0～1；Subjects underwent TURBT surgery or partial cystectomy and imaging diagnosis, which was determined to be muscular infiltrating urothelial carcinoma of the bladder (urothelial carcinoma being the main pathological component: 50%) and planned to undergo radical total cystectomy + lymph node dissection + urine flow diversion; cT2-T4a N0 M0 (CT/MRI ± PET/CT)；Undergo TURBT or partial cystectomy；Tissue examination specimens with TURBT or partial cystectomy；Expected survival ≥3 months；Immunohistochemical staining of tissue after final TURBT or partial cystectomy showed IHC 2+ or 3+；The major organs are functioning normally, the following criteria are met:

1. The blood routine examination criteria should meet (no blood transfusion and no treatment with granulocyte colony stimulating factor within 14 days before enrollment) :

   i. Absolute count of neutrophils (ANC) ≥1,000/mm3 ii. Platelet count ≥75,000/mm3 iii. Hemoglobin ≥ 8.0g /dL
2. Liver function:

   i. Total bilirubin ≤1.5× prescribed ULN or direct bilirubin ≤ULN for subjects with total bilirubin levels >1.5×ULN ii. Upper limit of normal values (ULN) ≤2.5 times of alanine Aminotransferase (ALT) and aspartate Aminotransferase (AST) Note: ≤1.5× ULN (This criterion only applies to patients who have not received anticoagulant therapy; Patients receiving anticoagulant therapy should keep anticoagulants within therapeutic limits);
3. Kidney function:

The Cockcroft-Gault formula was used to determine the creatinine clearance (CrCl) > 30 mL/min.

Subjects (or their legal representatives) must sign an informed consent form (ICF) indicating that they understand the purpose and procedures of the study and are willing to participate in the study; Fertile women must have a negative pregnancy test result (beta-hCG) (urine or serum) within 7 days before the study drug is first administered.

Exclusion criteria: Previously received anti-PD-1, anti-PD-L1, anti-PD-L2 therapy, including adjuvant therapy stage；Known allergy to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components；Those who had received other antitumor therapy (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks prior to study therapy, or had not recovered from previous toxicity (except for 2 degree hair loss and 1 degree neurotoxicity)；Pregnant or lactating woman；HIV positive；People with active hepatitis B or C；A history of definite active tuberculosis；Have active autoimmune diseases requiring systemic treatment within the past 2 years (e.g., use of disease-regulating drugs, corticosteroids, or immunosuppressive drugs) that allow for relevant replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for renal or pituitary insufficiency)；Other serious, uncontrolled concomitant diseases that may affect protocol adherence or interfere with interpretation of results, These include active opportunistic or progressive (severe) infections, uncontrolled diabetes, cardiovascular disease (heart failure of Grade Ⅲ or Ⅳ as defined by the New York Heart Association scale, heart block of degree Ⅱ or higher, myocardial infarction within the past 6 months, unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc.), or pulmonary disease (interstitial pneumonia, History of obstructive pulmonary disease and symptomatic bronchospasm)；Those who received the live vaccine within 4 weeks before treatment began；Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation；Major surgical procedures (excluding diagnostic surgery) within 4 weeks prior to the start of treatment；Those who have a history of psychotropic substance abuse and cannot abstain or have a history of mental disorders；A large amount of pleural fluid or ascites with clinical symptoms or symptomatic management；Have had other unhealed malignancies in the past 5 years, excluding those that are apparently cured or curable, such as basal or squamous cell skin cancer, localized low-risk prostate cancer, carcinoma in situ of the cervix or carcinoma in situ of the breast; Remarks: Patients with localized low-risk prostate cancer (defined as stage ≤T2b, Gleason score ≤7, and PSA≤20ng/mL at the time of prostate cancer diagnosis (as measured) who had received radical therapy and had no biochemical recurrence of prostate specific antigen (PSA) were eligible to participate in this study)；Urothelial carcinoma associated with upper urinary tract (renal pelvis and ureteral urothelial carcinoma)；Other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities that, according to the investigator, may increase the risks associated with study participation or may interfere with the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-13 (Estimated); Study Completion 2024-02-13 (Estimated)

PRIMARY OUTCOMES:
Safety | Up to 28 days
  Adverse events will be defined according to NCI CTCAE, Version 5.0

SECONDARY OUTCOMES:
Percent of Patients With Complete Response (CR) | Up to 3 months
  CR is defined by negative cystoscopy, urine cytology, and bladder biopsies.
Percent of Patients With Complete Response (CR) | Up to 12 months
  CR is defined by negative cystoscopy, urine cytology, and bladder biopsies.
Percent of Patients With Complete Response (CR) | Up to 24 months
  CR is defined by negative cystoscopy, urine cytology, and bladder biopsies.
1-yr and 2-yr Bladder-intact Event-free Survival (BI-EFS) | Up to 24 months
  Defined by time from enrollment to the occurrence of one of the following events: disease progression, switch to other therapy, intolerant adverse events, or death
Recurrence Free Survival (RFS) | Up to 24 months
  Defined by time from day of first treatment to recurrent NMIBC based on cystoscopy, cytology and/or biopsy.
Overall Survival (OS) | Up to 24 months
  Defined by time from day of first treatment to death
Cancer-Specific Survival | Up to 24 months
  Defined by time from day of first treatment to metastatic bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Haige Chen, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Jin D, Zang J, Qian L, Zhang T, Wu Y, Ding Y, Xie F, Tang H, Xia J, Cao D, Zhang R, Zhuang G, Chen H. Disitamab vedotin combined with toripalimab and radiotherapy for multimodal organ-sparing treatment of muscle invasive bladder cancer: a proof-of-concept study. Neoplasia. 2025 Oct;68:101216. doi: 10.1016/j.neo.2025.101216. Epub 2025 Aug 6. PMID 40774226